CLINICAL TRIAL: NCT05374148
Title: Respiratory Health Problems Among Workers in Ferrosilicon Alloys Industry in Aswan-Eygpt.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Bazied Dardir mohamed, Assistant lecturer, Assiut University
Other Study IDs: Respiratory ferrosilicon
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: health education — health education to prevent respiratory diseases among workers

SUMMARY:
To minimize the negative effects of exposure to silica, iron chips, and coke on the respiratory health of workers in the Ferro alloy factory, so it is important to assess and diagnose their health-related effects. Early reporting, diagnosis, and intervention can limit the severity of health hazards, improve health services. To our knowledge, no local previous studies were done in this area. All over the world there is no sufficient information relating to this industry and its health hazards.

DETAILED DESCRIPTION:
Ferrosilicon alloy is a mixture of iron and silicon. It's added to steel and cast iron. By oxidation of the iron, it offers superior properties to iron such as high strength, hardness, and resistance to corrosion and high temperatures. Around 90% of ferrosilicon alloys is consumed in the production of iron and steel. Silica dust is a secondary product of ferrosilicon industry. Its addition to concrete improve its chemical and physical properties[1] .

Ferrosilicon is an alloy of iron and silicon with high silicon content. Ferrosilicon alloys are produced in electric arc furnaces. At very high temperatures (2000°C). These furnaces are charged with quartz which is the main source of silica, iron chips, and coke which is used as a reducing agent. The industry process produces very fine particles of amorphous silica (SiO 2) powder(fume). The composition of the fumes varies somewhat according to which alloy is produced. In the production of ferrosilicon alloy with a high silicon content, the amount of Si02 in the fumes can be 80% or more[2].

Workers in the ferroalloy industry have been exposed to a variety of gases, fumes, and dust that may adversely affect the respiratory system. Among employees in Ferrosilicon plants, there is an increase in mortality rate from bronchitis, emphysema, and asthma[3]. Occupational exposure to respirable crystalline silica (SiO2) is one of the most common and serious hazards. It is considered a serious hazard for the ferrosilicon industry. Silicosis is the disease most associated with crystalline silica exposure. It causes by the inhalation of respirable crystalline silica dust [4]. It is a fibrotic lung disease progressive, irreversible, [5]. It is incurable but preventable[6]. Chronic Silicosis occurs due to the prolonged inhalation of respirable crystalline silica dust [4]. The major risk factors for developing silicosis include cumulative lifetime exposure, the total amount of inhaled crystalline Silica, silica size(0.5-3 µ) and individual susceptibility [6]. Thus, making silica dust one of the greater public health problems.

Silicosis is considered one of the most serious occupational diseases in the world. According to many previous studies, a large number of workers are exposed to silica dust throughout the world. At least 3.2 million workers in Europe and more than 2 million in the United States are exposed to silica dust[4] . In Asia, the prevalence of silicosis is up to 55% among workers exposed to silica dust, while in Latin America, the prevalence is up to 37%[8] In Egypt ,the prevalence rate of silicosis ranges from 18.5 % to 45.8% among workers exposed to free crystalline silica dust[9] Although many studies illustrated the relationship between silica exposure and silicosis occurrence in a different industries , there are no sufficient studies relating to the ferrosilicon industry and its respiratory hazards.

ELIGIBILITY:
Inclusion Criteria:

* Active working miners working in ferrosilicon alloy factory with minimum exposure 5 years.
* Workers exposed to silica, iron chips, and coke in quarry and Furnaces areas.
* Have free pre-employment records especially free chest x-rays. have no previous pre- employment history of any chest problems.

Exclusion Criteria:

* • Workers don't record silica, iron chips, and coke exposer as in the administration department.

  * Workers with less than 5-year exposure.
  * Workers are known to have chest diseases before joining the work for example emphysema and COPD.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: workers exposed to free silica who have a free pre-employment records
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
prevalence | 1 year
  prevalence of silicosis among ferrosilicon industry workers.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalliny MS, Bassyouni MI. Immune response due to silica exposure in Egyptian phosphate mines. J Health Care Poor Underserved. 2011;22(4 Suppl):91-109. doi: 10.1353/hpu.2011.0156. PMID 22102308
- [Background] Leung CC, Yu IT, Chen W. Silicosis. Lancet. 2012 May 26;379(9830):2008-18. doi: 10.1016/S0140-6736(12)60235-9. Epub 2012 Apr 24. PMID 22534002